CLINICAL TRIAL: NCT05639517
Title: The Effect of Augmented Reality Based Telerehabilitation Application on Neuromuscular and Sensorimotor Parameters in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-985
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients in this group will receive spinal stabilization training through augmented reality based telerehabilitation application.
  Interventions: Other: Augmented Reality Based Telerehabilitation Application
- Group 2 (Active Comparator): Patients in this group will receive spinal stabilization training face-to-face.
  Interventions: Other: Training face-to-face

INTERVENTIONS:
Other: Augmented Reality Based Telerehabilitation Application — Spinal stabilization training with augmented reality-based telerehabilitation will be applied twice a week for 8 weeks.
  Arms: Group 1
Other: Training face-to-face — Spinal stabilization training will be applied face-to-face twice a week for 8 weeks.
  Arms: Group 2

SUMMARY:
Core stability, which is affected from the early period in with patients Multiple Sclerosis (PwMS), is due to deterioration in the somatosensory, motor and musculoskeletal systems. Based on the knowledge that core stability is effective on many functions, it is seen that trunk stabilization exercises are included in the physiotherapy and rehabilitation programs of patients. However, the effectiveness of augmented reality-based telerehabilitation application, which includes trunk stabilization training in PwMS, has not been adequately investigated in the literature. The aim of the study is to investigate the effectiveness of augmented reality-based telerehabilitation application, which includes trunk stabilization training, on neuromuscular and sensorimotor parameters in PwMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relapsing remitting MS by a neurologist,
* Having a disability level between 1 and 5 according to the Expanded Disability Status Scale (EDSS),
* Those who get over 24 points in the Standardized Mini Mental State Test (SMMT),
* Those who have not had an MS attack in the last three months,
* Volunteer individuals

Exclusion Criteria:

* Receiving corticosteroid therapy in the last 4 weeks,
* Having additional neurological disease that may cause balance disorder
* Individuals who have had surgery related to the spine, hip, knee or ankle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Balance | Change from baseline at 8 weeks
  MiniBESTest will be used to evaluate the static and dynamic balance.It consists of 14 questions including antisipatuar postural reaction, reactive postural control, sensory orientation and dynamic balance. The test is scored between 0-28 points. The highest score indicates good balance.

SECONDARY OUTCOMES:
Muscle Activity | Change from baseline at 8 weeks
  An 8-channel superficial EMG system will be used to measure signals from the quadriceps and tibialis anterior muscles.Electrodes will be placed according to SENIAM criteria.The signals received from the muscles of the individuals will be recorded during standing up from sitting. As a result, the average muscle activations of the muscles during the activity will be numerically recorded in %MVIC.
Core Muscle Endurance-Trunk Flexor | Change from baseline at 8 weeks
  The trunk flexor test will be performed with the arms crossed over the thorax, the trunk at 60 degrees of flexion, and the knees and hips flexed to 90 degrees. The test will be finished when the participant is unable to maintain the position. The time will be recorded.As the time increases, the endurance decreases.
Core Muscle Endurance- Trunk Extansor | Change from baseline at 8 weeks
  The trunk extensor test will be performed in the prone position, with the pelvis, hips and knees fixed to the bed. The participant will be asked to cross his arms over his body and position his body horizontally. The test will be finished when the participant is unable to maintain the horizontal position. The time will be recorded. As the time increases, the endurance decreases.
Core Muscle Endurance- Side Bridge | Change from baseline at 8 weeks
  While the participants are in the side-lying position, they will raise their hips and align their bodies in a straight line by getting support from their feet and elbows. The time will be recorded by asking them to maintain the position as much as possible.As the time increases, the endurance decreases.
Trunk Position Sense | Change from baseline at 8 weeks
  Inclinometer will be positioned at spinous process of 1th thoracic vertebrae and 1 sacral during trunk position sense assessment. Subject will be retreated to neutral position and asked to come back taught position while eyes closed. Test will be repeated 3 times and angle of deviation from 30 degree flexion position will be recorded and the average of the results will be taken.As the deflection angle increases, the sense of position deteriorates. As the deflection angle increases, the sense of position deteriorates.
Spinal mobility | Change from baseline at 8 weeks
  Spinal Mouse device will be used to evaluate spinal mobility. Measurements will be made between the spinous process of the 7th cervical vertebra and approximately the level of the 3rd sacral vertebra. Maximum degrees of right-left lateral flexion in the frontal plane and maximum degrees of flexion-extension in the sagittal plane will be measured and recorded.As the degree increases, the deformity also increases.
Fatique-Fatigue Severity Scale | Change from baseline at 8 weeks
  The Fatigue Severity Scale, which rates the severity of fatigue symptoms, consists of questions expressing 9 different conditions.A high score indicates increased fatigue severity. Patients with a score of <4 will be considered "not tired", and patients with a score of >4 will be considered "tired".
Fatigue- Fatigue Impact Scale | Change from baseline at 8 weeks
  Each question ranges from 0 (no problem) to 4 (maximum problem) in the scale that evaluates cognitive status, physical condition and psychological status. High scores indicate fatigue.